CLINICAL TRIAL: NCT04582799
Title: Extra-Corporeal Carbon Dioxide Removal for Acute Decompensation of Chronic Obstructive Pulmonary Disease: A Randomized Clinical Trial (The ORION Study)
Brief Title: Extracorporeal CO2 Removal for Acute Decompensation of COPD
Acronym: ORION
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment, termination of funding.
Sponsor: University of Bologna (Other)
Collaborators: University of Milan (Other); University of Turin, Italy (Other); University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, V. Marco Ranieri, Full Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORION
Record Dates: First submitted 2020-10-03; First posted 2020-10-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; ECCO2R
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (NIV) (Active Comparator): Patients in the control group will be treated with non-invasive ventilation only.
  Interventions: Device: NIV
- Extracorporeal CO2 Removal (NIV+ECCO2R) (Experimental): Patients in the treatment group will be treated with non-invasive ventilation combined with Extracorporeal CO2 Removal.
  Interventions: Device: ECCO2R; Device: NIV

INTERVENTIONS:
Device: ECCO2R — Extracorporeal CO2 Removal
  Arms: Extracorporeal CO2 Removal (NIV+ECCO2R)
Device: NIV — Non-invasive ventilation

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of death worldwide, resulting in a social and economic burden that is substantial and increasing. Exacerbations affect the prognosis and quality of life of patients with COPD. Hospital mortality of patients admitted for a hypercapnic exacerbation of COPD is approximately 10% and the long-term outcome is poor. In addition, hypercapnic exacerbation of COPD have serious negative impacts on patient quality of life, lung function and costs. Thus, prompt treatment of exacerbations may impact the clinical progression of COPD by ameliorating quality of life and prognosis.

Standard of care for patients with COPD exacerbation that need ICU admission for management of acute hypercapnic respiratory failure and severe respiratory acidosis is non-invasive ventilation (NIV). When NIV fails (arterial pH remains < 7.30), invasive ventilation through endotracheal intubation is initiated to restore adequate gas-exchange. Extracorporeal circuits designed to remove CO2 (ECCO2R) may enhance the efficacy of NIV to remove CO2 and avoid the worsening of respiratory acidosis.

A recent matched cohort study with historical control, showed that: (a) the hazard of being intubated was three times higher in patients treated with "NIV-only" than in patients treated with "NIV-plus-ECCO2R"; (b) hospital mortality was significantly lower in "NIV plus ECCO2R" than in "NIV-only" [8% (95% CI 1.0-26.0%) vs. 33% (95% CI 18.0-57.5%), respectively]. However, ECCO2R-related complications were observed in almost half of the patients.

The consistency of the above discussed data, and the observation of the continuous increase use of ECCO2R despite the lack of solid evidence confirm that the equipoise regarding the use of ECCO2R may justify a randomized clinical trial to evaluate whether patients with respiratory acidosis refractory to NIV should be intubated and take the risks associated with invasive mechanical ventilation, or should be connected to ECCO2R to avoid intubation, but run the risk of the potentially serious ECCO2R-related complication The main objective of this randomized multicenter clinical trial is to test the hypothesis that in patients with acute life-threatening exacerbation of COPD, use of ECCO2R could increase event-free survival as compared to standard of care.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of death worldwide, resulting in a social and economic burden that is substantial and increasing. Exacerbations affect the prognosis and quality of life of patients with COPD. Hospital mortality of patients admitted for a hypercapnic exacerbation of COPD is approximately 10% and the long-term outcome is poor. In addition, hypercapnic exacerbation of COPD have serious negative impacts on patient quality of life, lung function and costs. Thus, prompt treatment of exacerbations may impact the clinical progression of COPD by ameliorating quality of life and prognosis.

The pathophysiological hallmarks of COPD patients include expiratory flow limitation and small airway closure. Under these circumstances, a prolonged expiratory time is the compensatory mechanism patients adopt to maintain a stable tidal breathing. COPD exacerbations result in higher respiratory rates and reduced expiratory time, leading to dynamic hyperinflation, elevated intrathoracic pressures, and excessive work of breathing. Alteration of the balance between (a) the decreased capacity of the respiratory muscles to generate pressure, and (b) the increased mechanical respiratory load due to expiratory flow limitation and small airway closure leads to CO2 retention. The consequent reduction of alveolar ventilation leads to a further worsening of CO2 retention and increased work of breathing. This vicious circle is the underlying mechanisms responsible of acute respiratory failure requiring admission in the intensive care unit (ICU) for ventilatory support.

Standard of care for patients with COPD exacerbation that need ICU admission for management of acute hypercapnic respiratory failure and severe respiratory acidosis is non-invasive ventilation (NIV). When NIV fails (arterial pH remains < 7.30), invasive ventilation through endotracheal intubation is initiated to restore adequate gas-exchange.

Extracorporeal circuits designed to remove CO2 (ECCO2R) have been used in patients with acute hypercapnic respiratory failure since ECCO2R may enhance the efficacy of NIV to remove CO2 and avoid the worsening of respiratory acidosis. Although available studies are limited to case series, several ECCO2R devices have been developed and proposed for the clinical use in patients with COPD. These systems often represent modifications of renal replacement therapy circuits, and are characterized by:

1. veno-venous by-pass systems
2. extracorporeal blood flow of 0.3-0.5 litres/min
3. 13 Fr bore catheters or a single co-axial catheter
4. very low doses or no heparin
5. minimal volumes for "priming"

This technological implementation of ECCO2-R is therefore closer to device for renal replacement therapy than full ECMO. CO2 is removed through a double-lumen catheter and constantly propelled, by a non-occlusive rotating pump, though an artificial membrane lung (a filter adding oxygen and removing carbon dioxide) connected to a source of 100% O2 (flow 6-8 liters/min). These systems are able to reduce PaCO2 by 20-25%.

A recent matched cohort study with historical control, compared "NIV-plus-ECCO2R" and "NIV-only" in patients at risk of NIV failure, and showed that (a) the hazard of being intubated was three times higher in patients treated with "NIV-only" than in patients treated with "NIV-plus-ECCO2R"; (b) hospital mortality was significantly lower in "NIV plus ECCO2R" than in "NIV-only" [8% (95% CI 1.0-26.0%) vs. 33% (95% CI 18.0-57.5%), respectively]. However, ECCO2R-related complications were observed in almost half of the patients. A recent systematic review evaluated the efficacy and safety of ECCO2R in patients with hypercapnic respiratory failure across 12 studies and showed that the majority of patients were either successfully weaned from mechanical ventilation or sustained on NIV, avoiding intubation. However, this high success rates, was associated with a high frequency of potentially severe complications.

The consistency of the above discussed data, and the observation of the continuous increase use of ECCO2R despite the lack of solid evidence confirm that the equipoise regarding the use of ECCO2R may justify a randomized clinical trial to evaluate whether patients with respiratory acidosis refractory to NIV should be intubated and take the risks associated with invasive mechanical ventilation, or should be connected to ECCO2R to avoid intubation, but run the risk of the potentially serious ECCO2R-related complication

Objectives:

The main objective of this randomized multicenter clinical trial is to test the hypothesis that in patients with acute life-threatening exacerbation of COPD, use of ECCO2R could increase event-free survival as compared to standard of care. Event free survival is defined as survival at day 28 free of any of the followings: (a) development of sepsis; (b) occurrence of a second episode of COPD exacerbation requiring or not mechanical ventilation; (c) occurrence of severe hypoxemia; (d) prolonged mechanical ventilation (e) death.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 and younger than 90 years
* Documented clinical history of COPD
* ICU admission for exacerbation of COPD requiring non-invasive ventilatory support After two hours of NIV at least two of the following criteria must be fulfilled
* arterial pH ≤ 7.25
* respiratory rate ≥30 breaths/min
* use of accessory muscles or paradoxical abdominal movements

Exclusion Criteria:

* mean arterial pressure <60 mmHg despite infusion of fluids and vasoactive drugs
* ratio of arterial-to-inspired oxygen O2 fraction (PaO2/FiO2) ≤ 150 with FiO2 of less than 0.6 and PEEP of at least 5 cm H2O
* contraindications to anticoagulation (i.e. any of the following: platelet count <50,000/mm3; prothrombin time-international normalized ratio (INR) >1.5; stroke or severe head trauma or intracranial arterio-venous malformation, or cerebral aneurysm, or central nervous system mass lesion within the previous 3 months; epidural catheter in place or expected to be positioned during the study; history of congenital bleeding diatheses; gastrointestinal bleeding within the 6 weeks prior to study entry; esophageal varices, chronic jaundice, cirrhosis, or chronic ascites; trauma);
* heparin-induced thrombocytopenia;
* body weight >120 Kg;
* contraindication to continuation of active treatment;
* failure to obtain consent
* catheter access to femoral vein or jugular vein impossible
* pneumothorax
* inclusion in other trials
* patient moribund
* severe liver insufficiency (Child-Pugh scores > 7) or fulminant hepatic failure
* diagnosed with acute or chronic neuromuscular disease
* required chronic mechanical ventilation prior to hospital admission

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Combined 28-day mortality or surrogate events | 28 days after enrollment
  Incidence of death, prolonged mechanical ventilation, development of septic shock, development of severe hypoxemia, second episode of COPD exacerbation

SECONDARY OUTCOMES:
Endotracheal intubation | 28 days after enrollment
  Cumulative incidence of endotracheal intubation
Tracheostomy | 28 days after enrollment
  Cumulative incidence of tracheostomy
Hospital length-of-stay | Whole hospital stay
  Duration of stay in the hospital
ICU length-of-stay | Whole ICU stay
  Duration of stay in the intensive care unit
90-day mortality | 90 days after enrollment
  Incidence of death

CONTACTS AND LOCATIONS:
Overall Officials: V. Marco Ranieri, M.D., Study Chair — University of Bologna; Stefano Nava, M.D., Study Chair — University of Bologna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tonetti T, Pisani L, Cavalli I, Vega ML, Maietti E, Filippini C, Nava S, Ranieri VM. Extracorporeal carbon dioxide removal for treatment of exacerbated chronic obstructive pulmonary disease (ORION): study protocol for a randomised controlled trial. Trials. 2021 Oct 19;22(1):718. doi: 10.1186/s13063-021-05692-w. PMID 34666820